CLINICAL TRIAL: NCT03921866
Title: Observational Cohort Study of Patients With Hormone Receptor-positive Metastatic Breast Cancer Treated With Palbociclib (Ibrance(Registered)) as Part of the United Kingdom Ibrance (Registered) Patient Program (IPP); the Real Outcomes Ibrance (Registered) Study (ROIS)
Brief Title: UK Ibrance Patient Program (IPP) Study
Acronym: ROIS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001194; ROIS (Other: Alias Study Number)
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-06

CONDITIONS: HR+/HER2- Locally Advanced, Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Palbociclib — Palbociclib

SUMMARY:
What are the real-world treatment patterns, patients' characteristics, clinical outcomes and healthcare resource utilisation associated with palbociclib treatment in the 3 years following initiation in United Kingdom patients with hormone receptor-positive, human epidermal growth factor 2-negative metastatic breast cancer treated as part of the IPP?

DETAILED DESCRIPTION:
Hormone receptor positive (HR+) breast cancer (BC) represents the largest therapeutic subtype of the disease, accounting for 60 to 65% of all malignant neoplasms of the breast. Palbociclib (Ibrance®) is a small-molecule inhibitor of cyclin-dependent kinases 4 and 6 (CDK4/6) which in clinical trial settings has been shown to increase progression-free survival (PFS) for patients with HR+, human epidermal growth factor 2-negative (HER2-) metastatic breast cancer (MBC). Palbociclib first received a European Union (EU) marketing authorisation in September 2016, to be commercialised as Ibrance® by Pfizer. Palbociclib was recommended for use with an aromatase inhibitor in patients with HR+/HER2- locally advanced and MBC in the National Health Service (NHS) in England by the National Institute for Health and Care Excellence (NICE) in November 2017 and by the Scottish Medicines Consortium (SMC) in December 2017. In order to provide access to palbociclib in the United Kingdom (UK) during the NICE/SMC appraisal period, the Ibrance® Patient Program (IPP) was initiated and run by Pfizer between April 2017 until a positive NICE/SMC appraisal in November 2017 (for England and Wales) or December 2017 (for Scotland).

Pfizer are interested in the opportunity to collect data from patients who received palbociclib as part of the UK IPP, to better understand patients' characteristics in a routine care setting, treatment persistence and dose management, clinical outcomes, and healthcare resource utilisation. This study will provide real-world evidence on patients' clinical progression and experience of treatment with palbociclib in routine clinical settings in a UK context.

Research question:

What are the real-world treatment patterns, patients' characteristics, clinical outcomes and healthcare resource utilisation associated with palbociclib treatment in the 3 years following initiation in United Kingdom patients with HR+/HER2- MBC treated as part of the IPP?

ELIGIBILITY:
Inclusion criteria:

All patients meeting the following eligibility criteria will be included in the study:

* Patients enrolled into the IPP at one of the selected hospitals (see Annex 1 for IPP enrolment letter).
* Patients who received ≥1 dose of palbociclib as part of the IPP at one of the selected sites.
* For sites where data collection is performed by pH Associates, written informed consent will be required from living patients to access their medical records.
* Patient aged ≥18 years old at enrollment into the IPP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women over the age of 18 who entered into the UK IPP
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United Kingdom (8):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Brighton Sussex Cancer Centre, Brighton
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guys and St Thomas' NHS Trust, London
  - Maidstone Hospital, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge, Metropolitan Borough of Wirral
  - Newcastle Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Palmieri C, Musson A, Harper-Wynne C, Wheatley D, Bertelli G, Macpherson IR, Nathan M, McDowall E, Bhojwani A, Verrill M, Eva J, Doody C, Chowdhury R. A real-world study of the first use of palbociclib for the treatment of advanced breast cancer within the UK National Health Service as part of the novel Ibrance(R) Patient Program. Br J Cancer. 2023 Sep;129(5):852-860. doi: 10.1038/s41416-023-02352-5. Epub 2023 Jul 19. PMID 37468569
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had hormone receptor (HR) positive, human epidermal growth factor 2 (HER2) negative metastatic breast cancer (MBC) and were treated with palbociclib in the United Kingdom Ibrance Patient Program (IPP), in between 2018 to 2021 were observed in this study. Data collected from hospital medical records were observed both retrospectively and prospectively for approximately 3 years in this study.
Groups:
- Palbociclib: Participants with HR positive/HER2 negative MBC who received at least 1 dose of palbociclib as part of the IPP were observed during the study. Data was collected both retrospectively and prospectively, from participants' medical records for a maximum of 3 years following index date. Index date was defined as the palbociclib treatment initiation date.
Period: Overall Study
Arm/Group | Palbociclib
Started | 191
Completed | 191 (Out of these 191 participants, 3 participants died. But data available before censoring date for these 3 participants were observed and included in results.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study.
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Due to low enrollment in one category, providing data would risk re-identification of participants.
  Male | NA — Due to low enrollment in one category, providing data would risk re-identification of participants.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 169
  Black | 8
  Asian | 1
  Other | 1
  Missing | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants According to Treatment Lines
Description: Percentage of participants according to treatment lines during anytime between breast cancer (BC) diagnosis and index date were reported in this outcome measure. Treatment lines included: 1) 1st line where, palbociclib was prescribed as the first line treatment for MBC, 2) 1st line palbociclib added to letrozole where, palbociclib was prescribed as the first line treatment along with ongoing letrozole treatment which was prescribed more than 3 months prior to initiation of palbociclib, 3) 2nd line where palbociclib was prescribed as the second or later treatment line for MBC.
Time Frame: At baseline
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  1st Line | 72
  1st Line palbociclib added to letrozole | 16
  2nd Line | 10
  Unclassified | 2

2. Primary Outcome: Time From Letrozole to Palbociclib Initiation
Description: Time from letrozole was defined as duration from the start date of letrozole which was ongoing at the time of palbociclib treatment initiation up to the index date.
Time Frame: At baseline
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Palbociclib
Number analyzed (Participants) | 25
Days | 430.8 (770.8)

3. Primary Outcome: Number of Participants With Menopausal Status
Description: Number of participants with menopausal status as pre-menopausal, peri-menopausal, post-menopausal and not applicable (NA), during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here "number analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants
  At initial diagnosis: Pre-menopausal | 86
  At initial diagnosis: Post-menopausal | 94
  At initial diagnosis: Peri-menopausal | 6
  At initial diagnosis: NA | 1
  At initial diagnosis: Missing | 4
  At recurrence of disease: Pre-menopausal: number analyzed (Participants) | 134
  At recurrence of disease: Pre-menopausal | 35
  At recurrence of disease: Post-menopausal: number analyzed (Participants) | 134
  At recurrence of disease: Post-menopausal | 94
  At recurrence of disease: Peri-menopausal: number analyzed (Participants) | 134
  At recurrence of disease: Peri-menopausal | 5
  Metastatic setting: Pre-menopausal | 55
  Metastatic setting: Post-menopausal | 127
  Metastatic setting: Peri-menopausal | 8
  Metastatic setting: NA | 1

4. Primary Outcome: Percentage of Participants According to Disease Free Interval at Palbociclib Initiation
Description: Disease free interval was defined as the time from the date of last known neo-adjuvant hormone therapy to the date of MBC diagnosis.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 166
Percentage of participants
  More than 12 months | 29
  Less than or equal to (<=)12 months | 37
  De novo metastatic disease | 34

5. Primary Outcome: Percentage of Participants With Primary or Recurrent Metastatic Breast Cancer Diagnosis
Description: Percentage of participants with de novo and recurrent metastatic disease, during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Participants with de novo metastatic disease | 30
  Participants with recurrent disease | 70

6. Primary Outcome: Percentage of Participants With Lymph Nodes Involvement
Description: Percentage of participants with lymph nodes involvement during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. Data for this outcome measure is also presented by de novo status.
Time Frame: At baseline
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies number of participants evaluable for specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 188
Percentage of participants
  Initial diagnosis | 58
  De novo metastatic: number analyzed (Participants) | 55
  De novo metastatic | 58
  Non de novo metastatic: number analyzed (Participants) | 133
  Non de novo metastatic | 58

7. Primary Outcome: Number of Lymph Nodes Involved
Description: Number of lymph nodes involved during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. Data for this outcome measure is also presented by de novo status.
Time Frame: At baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Lymph nodes
Arm/Group | Palbociclib
Number analyzed (Participants) | 96
Lymph nodes
  Initial diagnosis | 4.4 (4.4)
  De novo metastatic: number analyzed (Participants) | 24
  De novo metastatic | 4.4 (3)
  Non de novo metastatic: number analyzed (Participants) | 72
  Non de novo metastatic | 4.4 (4.8)

8. Primary Outcome: Number of Participants With Estrogen, Progesterone and Human Epidermal Growth Factor 2 (HER2) Receptor Status
Description: Number of participants with estrogen, progesterone and HER2 receptor status during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, "number analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants
  Estrogen receptor status at initial diagnosis: Positive | 178
  Estrogen receptor status at initial diagnosis: Negative | 2
  Estrogen receptor status at initial diagnosis: Missing | 11
  HER2 receptor status at initial diagnosis: Positive | 1
  HER2 receptor status at initial diagnosis: Negative | 170
  HER2 receptor status at initial diagnosis: Missing | 20
  Progesterone receptor status at initial diagnosis: Positive | 38
  Progesterone receptor status at initial diagnosis: Negative | 25
  Progesterone receptor status at initial diagnosis: Not known | 14
  Progesterone receptor status at initial diagnosis: Missing | 114
  Estrogen receptor status at recurrence of disease: Positive: number analyzed (Participants) | 77
  Estrogen receptor status at recurrence of disease: Positive | 73
  Estrogen receptor status at recurrence of disease: Negative: number analyzed (Participants) | 77
  Estrogen receptor status at recurrence of disease: Negative | 2
  Estrogen receptor status at recurrence of disease: Missing: number analyzed (Participants) | 77
  Estrogen receptor status at recurrence of disease: Missing | 2
  HER2 receptor status at recurrence of disease: Negative: number analyzed (Participants) | 77
  HER2 receptor status at recurrence of disease: Negative | 75
  HER2 receptor status at recurrence of disease: Missing: number analyzed (Participants) | 77
  HER2 receptor status at recurrence of disease: Missing | 2
  Progesterone receptor status at recurrence of disease: Positive: number analyzed (Participants) | 134
  Progesterone receptor status at recurrence of disease: Positive | 38
  Progesterone receptor status at recurrence of disease: Negative: number analyzed (Participants) | 134
  Progesterone receptor status at recurrence of disease: Negative | 25
  Progesterone receptor status at recurrence of disease: Not known: number analyzed (Participants) | 134
  Progesterone receptor status at recurrence of disease: Not known | 14
  Progesterone receptor status at recurrence of disease: Missing: number analyzed (Participants) | 134
  Progesterone receptor status at recurrence of disease: Missing | 57
  Estrogen receptor status at metastatic setting: Positive | 130
  Estrogen receptor status at metastatic setting: Negative | 2
  Estrogen receptor status at metastatic setting: No rebiopsy in metastatic setting | 50
  Estrogen receptor status at metastatic setting: Missing | 9
  HER2 receptor status at metastatic setting: Negative | 131
  HER2 receptor status at metastatic setting: No rebiopsy in metastatic setting | 50
  HER2 receptor status at metastatic setting: Missing | 10
  Progesterone receptor status at metastatic setting: Positive: number analyzed (Participants) | 134
  Progesterone receptor status at metastatic setting: Positive | 76
  Progesterone receptor status at metastatic setting: Negative: number analyzed (Participants) | 134
  Progesterone receptor status at metastatic setting: Negative | 35
  Progesterone receptor status at metastatic setting: Not known: number analyzed (Participants) | 134
  Progesterone receptor status at metastatic setting: Not known | 22
  Progesterone receptor status at metastatic setting: Missing: number analyzed (Participants) | 134
  Progesterone receptor status at metastatic setting: Missing | 1

9. Primary Outcome: Percentage of Participants Who Had Rebiopsy After Metastatic Disease Diagnosis
Description: Percentage of participants who had rebiopsy during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 127
Percentage of participants | 61

10. Primary Outcome: Percentage of Participants According to Tumor Stage
Description: Percentage of participants with tumor stages 0, 1, 2, 3 and 4, as per Tumor, Node, Metastasis (TNM) staging system, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. As per TNM staging system, tumor stage 0 indicates main tumor cannot be found; tumor stages 1, 2, 3 and 4 refers to the size and/or extent of the main tumor. The higher the number, the larger the tumor and/or the more it has spread into nearby tissues. Data for this outcome measure is also presented by de novo status.
Time Frame: At baseline
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 160
Percentage of participants
  At initial diagnosis: Stage 0 | 5
  At initial diagnosis: Stage 1 | 19
  At initial diagnosis: Stage 2 | 51
  At initial diagnosis: Stage 3 | 21
  At initial diagnosis: Stage 4 | 4
  De novo metastatic: Stage 0: number analyzed (Participants) | 49
  De novo metastatic: Stage 0 | 12
  De novo metastatic: Stage 1: number analyzed (Participants) | 49
  De novo metastatic: Stage 1 | 8
  De novo metastatic: Stage 2: number analyzed (Participants) | 49
  De novo metastatic: Stage 2 | 39
  De novo metastatic: Stage 3: number analyzed (Participants) | 49
  De novo metastatic: Stage 3 | 29
  De novo metastatic: Stage 4: number analyzed (Participants) | 49
  De novo metastatic: Stage 4 | 12
  Non de novo metastatic: Stage 0: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 0 | 2
  Non de novo metastatic: Stage 1: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 1 | 23
  Non de novo metastatic: Stage 2: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 2 | 56
  Non de novo metastatic: Stage 3: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 3 | 18
  Non de novo metastatic: Stage 4: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 4 | 1

11. Primary Outcome: Percentage of Participants According to Nodal Status
Description: Percentage of participants with nodal stages 0, 1, 2 and 3, as per TNM staging system, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. As per TNM staging system, nodal stage 0 indicates no cancer in regional lymph nodes; nodal stages 1= cancer has spread to 1 to 3 lymph nodes; nodal stage 2= cancer has spread to 4 to 9 lymph nodes, nodal stage 3= indicates the cancer has spread to 10 or more lymph nodes. Data for this outcome measure is also presented by de novo status.
Time Frame: At baseline
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 157
Percentage of participants
  At initial diagnosis: Stage 0 | 39
  At initial diagnosis: Stage 1 | 38
  At initial diagnosis: Stage 2 | 11
  At initial diagnosis: Stage 3 | 12
  De novo metastatic: Stage 0: number analyzed (Participants) | 46
  De novo metastatic: Stage 0 | 35
  De novo metastatic: Stage 1: number analyzed (Participants) | 46
  De novo metastatic: Stage 1 | 30
  De novo metastatic: Stage 2: number analyzed (Participants) | 46
  De novo metastatic: Stage 2 | 15
  De novo metastatic: Stage 3: number analyzed (Participants) | 46
  De novo metastatic: Stage 3 | 20
  Non de novo metastatic: Stage 0: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 0 | 41
  Non de novo metastatic: Stage 1: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 1 | 41
  Non de novo metastatic: Stage 2: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 2 | 9
  Non de novo metastatic: Stage 3: number analyzed (Participants) | 111
  Non de novo metastatic: Stage 3 | 9

12. Primary Outcome: Percentage of Participants According to Metastasis
Description: Percentage of participants with metastasis stages 0 and 1, as per TNM staging system, during anytime between MBC disease diagnosis and index date were reported in this outcome measure. As per TNM staging system, metastasis stage 0 indicates cancer has not spread to other parts of the body; metastasis stage 1 indicates that the cancer has spread to distant parts of the body. Data for this outcome measure is also presented by de novo status.
Time Frame: At baseline
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 174
Percentage of participants
  At initial diagnosis: Stage 0 | 64
  At initial diagnosis: Stage 1 | 36
  De novo metastatic: Stage 1: number analyzed (Participants) | 57
  De novo metastatic: Stage 1 | 100
  Non de novo metastatic: Stage 0: number analyzed (Participants) | 117
  Non de novo metastatic: Stage 0 | 96
  Non de novo metastatic: Stage 1: number analyzed (Participants) | 117
  Non de novo metastatic: Stage 1 | 4

13. Primary Outcome: Tumor Size at Palbociclib Initiation
Time Frame: At baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Palbociclib
Number analyzed (Participants) | 162
Millimeters
  At Initial diagnosis | 35.4 (27.5)
  De novo metastatic status: number analyzed (Participants) | 48
  De novo metastatic status | 40.9 (36)
  Non de novo metastatic status: number analyzed (Participants) | 114
  Non de novo metastatic status | 33.1 (22.9)

14. Primary Outcome: Percentage of Participants According to Tumor Grade
Description: Percentage of participants with tumor grades, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. Grades of disease was classified as grades 1, 2 and 3. As per TNM system, grade 1= well differentiated cells, low grade; grade 2= moderately differentiated cells, intermediate grade and grade 3= poorly differentiated cells, high grade.
Time Frame: At baseline
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 170
Percentage of participants
  At initial diagnosis: Grade 1 | 10
  At initial diagnosis: Grade 2 | 56
  At initial diagnosis: Grade 3 | 34
  De novo metastatic: Grade 1: number analyzed (Participants) | 49
  De novo metastatic: Grade 1 | 4
  De novo metastatic: Grade 2: number analyzed (Participants) | 49
  De novo metastatic: Grade 2 | 63
  De novo metastatic: Grade 3: number analyzed (Participants) | 49
  De novo metastatic: Grade 3 | 33
  Non de novo metastatic: Grade 1: number analyzed (Participants) | 121
  Non de novo metastatic: Grade 1 | 12
  Non de novo metastatic: Grade 2: number analyzed (Participants) | 121
  Non de novo metastatic: Grade 2 | 53
  Non de novo metastatic: Grade 3: number analyzed (Participants) | 121
  Non de novo metastatic: Grade 3 | 35

15. Primary Outcome: Percentage of Participants With Ki-67 Protein Proliferation Index Recorded
Description: Percentage of participants with Ki-67 protein proliferation index during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. The Ki-67 protein is a cellular marker for proliferation. Ki-67 is a protein in cells that increases as cells prepare to divide into new cells. A staining process can measure the percentage of tumor cells that are positive for Ki-67. More positive cells hasten in dividing and forming new cells. Proliferation index was measured by the percentage of cells staining for Ki-67.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 173
Percentage of participants | 14

16. Primary Outcome: Ki-67 Protein Proliferation Index
Description: The Ki-67 protein is a cellular marker for proliferation. Ki-67 is a protein in cells that increases as cells prepare to divide into new cells. A staining process can measure the percentage of tumor cells that are positive for Ki-67. More positive cells hasten in dividing and forming new cells. Proliferation index was measured by the percentage of cells staining for Ki-67.
Time Frame: At baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of cells staining for Ki-67
Arm/Group | Palbociclib
Number analyzed (Participants) | 25
Percentage of cells staining for Ki-67 | 30.8 (23)

17. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Score (ECOG PS)
Description: ECOG PS measured quality of life of cancer participants on a 0 to 5 scale; 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity, ambulatory, able to carry out light/sedentary work; 2= ambulatory, capable of all self-care, unable to carry out any work activity, up >50 % of waking hours; 3= capable of only limited self-care, confined to bed/ chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5= dead. Higher scores indicated worsening of quality of life.
Time Frame: At baseline
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 112
Percentage of participants
  At initial diagnosis: Score 0: number analyzed (Participants) | 93
  At initial diagnosis: Score 0 | 68
  At initial diagnosis: Score 1: number analyzed (Participants) | 93
  At initial diagnosis: Score 1 | 25
  At initial diagnosis: Score 2: number analyzed (Participants) | 93
  At initial diagnosis: Score 2 | 8
  At recurrence of disease: Score 0: number analyzed (Participants) | 67
  At recurrence of disease: Score 0 | 45
  At recurrence of disease: Score1: number analyzed (Participants) | 67
  At recurrence of disease: Score1 | 40
  At recurrence of disease: Score 2: number analyzed (Participants) | 67
  At recurrence of disease: Score 2 | 15
  At metastatic diagnosis: Score 0 | 55
  At metastatic diagnosis: Score1 | 32
  At metastatic diagnosis: Score 2 | 12

18. Primary Outcome: Percentage of Participants With Recurrence Type
Description: Percentage of participants with recurrence type during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 127
Percentage of participants
  Distant | 77
  Locoregional | 23

19. Primary Outcome: Percentage of Participants According to Number of Metastatic Sites
Description: Percentage of participants according to number of metastatic sites during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 146
Percentage of participants
  1 | 45
  2 | 36
  3 | 14
  4 or more | 5

20. Primary Outcome: Percentage of Participants According to Location of Metastases
Description: Percentage of participants according to location of metastases, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 189
Percentage of participants
  Non-visceral | 67
  Visceral | 33

21. Primary Outcome: Percentage of Participants With Non-Visceral Location of Metastases
Description: Percentage of participants with non-visceral location of metastases, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 127
Percentage of participants
  Bone only metastases | 67
  Other non-visceral | 33

22. Primary Outcome: Number of Participants According to Metastatic Sites With Locoregional Recurrence
Description: Number of participants according to metastatic sites with locoregional recurrence, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. Metastatic sites with locoregional recurrence included bone, breast, lung, pleural, regional lymph nodes and other sites.
Time Frame: At baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 29
Participants
  Bone | 5
  Breast | 3
  Lung | 2
  Pleural | 1
  Regional lymph nodes | 2
  Other sites | 16

23. Primary Outcome: Duration of Disease at Initiation of Palbociclib
Description: Duration of BC disease was the time duration between date of BC disease diagnosis to palbociclib treatment initiation date.
Time Frame: At baseline
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 190
Months | 225.9 [1.9 to 1722.4]

24. Primary Outcome: Percentage of Participants Who Received Chemotherapy in Adjuvant or Neoadjuvant Setting
Description: Percentage of participants who received chemotherapy in adjuvant or neoadjuvant setting, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 46

25. Primary Outcome: Percentage of Participants Who Received Chemotherapy in Advanced, Disease Modifying or Metastatic Setting
Description: Percentage of participants who received chemotherapy in advanced, disease modifying or metastatic setting, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 15

26. Primary Outcome: Number of Lines of Prior Chemotherapy for Metastatic Disease
Description: Number of lines of prior chemotherapy for metastatic disease during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Chemotherapy lines
Arm/Group | Palbociclib
Number analyzed (Participants) | 29
Chemotherapy lines | 1.4 (0.7)

27. Primary Outcome: Percentage of Participants Who Received Luteinizing Hormone Releasing Hormone (LHRH) or Chemotherapy
Description: Percentage of participants who received LHRH or chemotherapy, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 53
Percentage of participants | 96

28. Primary Outcome: Percentage of Participants Who Received Endocrine Therapy in Adjuvant or Neoadjuvant Setting
Description: Percentage of participants who received endocrine therapy in adjuvant or neoadjuvant setting, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 61

29. Primary Outcome: Number of Participants With Types of Endocrine Therapy in Adjuvant or Neoadjuvant Setting
Description: Number of participants with types of endocrine therapy in adjuvant or neoadjuvant setting, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 137
Participants
  Adjuvant endocrine therapy: Anastrozole | 19
  Adjuvant endocrine therapy: Exemestane | 11
  Adjuvant endocrine therapy: Letrozole | 16
  Adjuvant endocrine therapy: Tamoxifen | 86
  Adjuvant endocrine therapy: Other | 5
  Neoadjuvant endocrine therapy: Anastrozole: number analyzed (Participants) | 7
  Neoadjuvant endocrine therapy: Anastrozole | 2
  Neoadjuvant endocrine therapy: Letrozole: number analyzed (Participants) | 7
  Neoadjuvant endocrine therapy: Letrozole | 2
  Neoadjuvant endocrine therapy: Tamoxifen: number analyzed (Participants) | 7
  Neoadjuvant endocrine therapy: Tamoxifen | 3

30. Primary Outcome: Percentage of Participants Who Received Endocrine Therapy in Advanced, Disease Modifying or Metastatic Setting
Description: Percentage of participants who received endocrine therapy in advanced, disease modifying or metastatic setting, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 38

31. Primary Outcome: Percentage of Participants With Type of Endocrine Therapy in Advanced, Disease Modifying or Metastatic Setting
Description: Percentage of participants with type of endocrine therapy in advanced, disease modifying or metastatic setting, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 99
Percentage of participants
  Anastrozole | 4
  Exemestane | 13
  Fulvestrant | 3
  Letrozole | 54
  Other | 12
  Tamoxifen | 14

32. Primary Outcome: Number of Lines of Prior Endocrine Therapy for Metastatic Disease
Description: Number of lines of prior endocrine therapy for metastatic disease during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Endocrine therapy lines
Arm/Group | Palbociclib
Number analyzed (Participants) | 73
Endocrine therapy lines | 1.4 (0.6)

33. Primary Outcome: Number of Participants Who Received Radiotherapy in Advanced, Disease Modifying or Metastatic Setting
Description: Number of participants who received radiotherapy in advanced, disease modifying or metastatic setting, during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants | 53

34. Primary Outcome: Percentage of Participants Who Received Concomitant Medications
Description: Percentage of participants who received concomitant medications, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 100

35. Primary Outcome: Number of Participants With Concomitant Medications Prescribed Along With Goserelin
Description: Number of participants with concomitant medications prescribed along with goserelin, during anytime between initial BC disease diagnosis and index date were reported in this outcome measure. Goserelin is the generic drug with a brand name Zoladex.
Time Frame: At baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 17
Participants
  Zoladex and Anastrozole | 1
  Zoladex and Letrozole | 10
  Zoladex and Tamoxifen then Exemestane | 1
  Zoladex only | 4
  Zoladex, Exemestane, Letrozole and Tamoxifen | 1

36. Primary Outcome: Number of Participants According to Number of Prior Treatments in Metastatic Setting
Description: Number of participants according to number of prior treatments in metastatic setting, during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants
  0 | 83
  1 | 58
  2 | 24
  3 | 12
  4 | 7
  5 | 4
  6 | 1
  8 | 1
  10 | 1

37. Primary Outcome: Number of Participants According to Number of Prior Chemotherapy and Hormone Therapy in Metastatic Setting
Description: Number of participants according to number of prior chemotherapy and hormone therapy in metastatic setting, during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants
  0 | 108
  1 | 46
  2 | 24
  3 | 6
  4 | 6
  5 | 1

38. Primary Outcome: Number of Participants According to Number of Prior Chemotherapies in Metastatic Setting
Description: Number of participants according to number of prior chemotherapies in metastatic setting, during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants
  0 | 162
  1 | 19
  2 | 7
  3 | 3

39. Primary Outcome: Number of Participants According to Number of Prior Hormone Therapies in Metastatic Setting
Description: Number of participants according to number of prior hormone therapies in metastatic setting, during anytime between MBC disease diagnosis and index date were reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Participants
  0 | 118
  1 | 52
  2 | 17
  3 | 3
  4 | 1

40. Secondary Outcome: Percentage of Participants With Their Starting Dose of Palbociclib
Description: Percentage of participants with their starting dose of palbociclib were reported.
Time Frame: Data collected at index date (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  125 milligrams (mg)/day | 97
  100 mg/day | 3

41. Secondary Outcome: Percentage of Participants Who Received Endocrine Therapy Along With Palbociclib
Description: Percentage of participants who received endocrine therapy along with palbociclib were reported in this outcome measure. Endocrine therapy includes anastrozole, exemestane, fulvestrant and letrozole.
Time Frame: Data collected from index date until lost to follow up or end of follow up, whichever occurred first (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 190
Percentage of participants
  Anastrozole | 3
  Exemestane | 7
  Fulvestrant | 1
  Letrozole | 89

42. Secondary Outcome: Percentage of Participants With Dose Reductions and Treatment Discontinuation
Description: Percentage of participants with dose reductions and treatment discontinuation were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Dose reduction | 41
  Treatment discontinuation | 54

43. Secondary Outcome: Number of Participants With Reasons for Palbociclib Discontinuation
Description: Number of participants with reasons for palbociclib discontinuation were reported in this outcome measure. Disease progression (PD) was defined as greater than or equal to (>=)20 percent (%) increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 millimeter (mm) or appearance of 1 or more new lesions. Adverse drug reactions (ADR) were defined as unintended, harmful events attributed to the use of drug. As per World Health Organisation (WHO) criteria for hematologic and nonhematologic toxicity grade 3 was defined as the severe/worst grade.
Time Frame: as for outcome 41
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 103
Participants
  Adverse drug reaction | 3
  Hematologic toxicity: Grade 3 | 1
  Non-hematologic: Grade 3 | 1
  Progression of disease | 83
  Other | 15

44. Secondary Outcome: Percentage of Participants With Temporary Discontinuation
Description: Percentage of participants with temporary discontinuation of palbociclib were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 40

45. Secondary Outcome: Percentage of Participants According to Time to Dose Reduction in First Line Therapy
Description: Percentage of participants according to time to dose reduction after palbociclib initiation in 1st line therapy were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 137
Percentage of participants
  Within 3 months | 19
  Between 3 to 6 months | 11
  Over 6 months | 12

46. Secondary Outcome: Time to Palbociclib Discontinuation
Description: Time to palbociclib discontinuation were observed in participants who permanently discontinued palbociclib and were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 103
Months | 8.3 [0.1 to 24.0]

47. Secondary Outcome: Number of Participants With First 3 Lines of Treatment After Progression
Description: Number of participants according to lines of treatment after progression were reported in this outcome measure.
Time Frame: Data collected from date of progression until lost to follow up or end of follow up period, whichever occurred first (for a maximum period of 3 years)
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies number of participants evaluable for specified rows. Participant can be included in more than 1 category.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 103
Participants
  1st line treatment | 80
  2nd line treatment: number analyzed (Participants) | 80
  2nd line treatment | 42
  3rd line treatment: number analyzed (Participants) | 42
  3rd line treatment | 20

48. Secondary Outcome: Doses Prescribed for First 3 Lines of Treatment After Progression
Description: Doses of drugs prescribed for first 3 lines of treatment after progression were reported in this outcome measure.
Time Frame: as for outcome 47
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Palbociclib
Number analyzed (Participants) | 79
Milligrams
  1st line - dose prescribed | 909.4 (1170.4)
  2nd line - dose prescribed: number analyzed (Participants) | 42
  2nd line - dose prescribed | 560.6 (1014.1)
  3rd line - dose prescribed: number analyzed (Participants) | 20
  3rd line - dose prescribed | 362.4 (531.0)

49. Secondary Outcome: Duration of First 3 Lines of Treatment After Progression
Description: Time duration of first 3 lines of treatment after progression up to lost to follow up or end of follow up period, whichever occurred first were reported in this outcome measure.
Time Frame: as for outcome 47
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Median (Full Range); unit: Days
Arm/Group | Palbociclib
Number analyzed (Participants) | 59
Days
  1st line treatment | 77.0 [0.0 to 592.0]
  2nd line treatment: number analyzed (Participants) | 33
  2nd line treatment | 67.0 [0.0 to 304.0]
  3rd line treatment: number analyzed (Participants) | 13
  3rd line treatment | 42 [0.0 to 91.0]

50. Secondary Outcome: Number of Completed Cycles of Palbociclib
Description: Number of 28-day cycles completed for palbociclib treatment were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Cycles | 15.0 (8.8)

51. Secondary Outcome: Percentage of Participants Who Received Letrozole and Fulvestrant With Palbociclib
Description: Percentage of participants who received letrozole and fulvestrant along with palbociclib were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 190
Percentage of participants
  Letrozole | 89
  Fulvestrant | 1

52. Secondary Outcome: Percentage of Participants With Progression Free Survival Following Palbociclib Initiation
Description: Progression free survival (PFS) was defined as the time from the index date to the date of first documented disease progression (PD) or death. PD was defined as >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions. Percentage of participants with progression free survival after index date were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 53

53. Secondary Outcome: Percentage of Participants Alive Following Palbociclib Initiation
Description: Percentage of participants who were alive after palbociclib initiation were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 71

54. Secondary Outcome: Percentage of Participants With Partial Response (PR) and Complete Response (CR) Following Palbociclib Initiation
Description: CR was defined as disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures less than (<)10 mm; PR was defined as >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Complete response | 2
  Partial response | 40

55. Secondary Outcome: Percentage of Participants With Stable Disease (SD) Following Palbociclib Initiation
Description: SD was defined as neither shrinkage for CR or PR nor increase for PD taking as reference smallest sum of longest diameters since treatment start. Alive participants with no events were censored at date of last response assessment. CR: disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures <10 mm; PR: >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 48

56. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the index date to the date of first documented PD or death. PD was defined as at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From index date to PD or death whichever occurred first (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Months | 19.5 [14.5 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated due to insufficient number of participants with events.

57. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the index date and the date of death from any cause. Participants who were still alive at the last date of data collection were censored.
Time Frame: From index date until date of death or date of censoring (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 190
Months | NA [NA to NA] — Median and 95% CI could not be calculated due to less number of participants with event.

58. Secondary Outcome: Time to Achieving Best Overall Response (BOR)
Description: Time to achieving BOR: time from index date until achievement of BOR: CR or PR, if CR was not achieved during follow-up. CR: disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures <10 mm; PR: >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm. Appearance of 1 or more new lesions; Alive participants with no events were censored at date of last response assessment.
Time Frame: From index date till date of BOR or date of censoring (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 185
Months | 3.5 [0.1 to 23.8]

59. Secondary Outcome: Duration of Follow-up Period
Description: Duration of follow-up period defined as the duration from index date until lost to follow up or end of follow up period, whichever occurred first, were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 190
Months | 20.8 (6)

60. Secondary Outcome: Percentage of Participants With Best Response (BR), Progressive Disease (PD) and Stable Disease (SD) to Palbociclib
Description: Percentage of participants with BR, PD and SD to palbociclib were reported in this outcome measure. BR was recorded for CR or PR. CR: disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures <10 mm; PR: >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions. SD: neither shrinkage for CR/PR nor increase for PD taking as reference smallest sum of longest diameters since treatment start. Alive participants with no events were censored at date of last response assessment.
Time Frame: From index date till BR (CR or PR, whichever occurred first), SD, PD or date of censoring (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Overall: CR | 2
  Overall: PR | 40
  Overall: PD | 7
  Overall: SD | 48
  De novo status: CR | 2
  De novo status: PR | 40
  De novo status: PD | 7
  De novo status: SD | 48
  Relapse status: CR | 2
  Relapse status: PR | 40
  Relapse status: PD | 7
  Relapse status: SD | 48

61. Secondary Outcome: Time to Best Response (BR)
Description: Time to BR: time from index date until achievement of BR:CR or PR, if CR not achieved during follow-up. CR: disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures <10 mm; PR: >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions. Alive participants with no events were censored at date of last response assessment. Data is also presented by de novo status and relapse status.
Time Frame: From index date till BR or date of censoring (for a maximum period of 3 years)
Population: as for outcome 6
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 185
Months
  Overall | 3.5 [0.1 to 23.8]
  De novo status: Metastatic disease: number analyzed (Participants) | 55
  De novo status: Metastatic disease | 3.4 [0.1 to 19.7]
  De novo status: Recurrent disease: number analyzed (Participants) | 130
  De novo status: Recurrent disease | 3.6 [0.2 to 23.8]
  Relapse status: More than 12 months: number analyzed (Participants) | 46
  Relapse status: More than 12 months | 3.9 [1.0 to 23.2]
  Relapse status: De novo metastatic disease: number analyzed (Participants) | 55
  Relapse status: De novo metastatic disease | 3.4 [0.1 to 19.7]
  Relapse status: <=12 months: number analyzed (Participants) | 59
  Relapse status: <=12 months | 3.8 [0.2 to 23.8]
  Relapse status: Missing: number analyzed (Participants) | 25
  Relapse status: Missing | 3.4 [0.3 to 11.0]

62. Secondary Outcome: Time to First Response
Description: Time to first response: time from index date until achievement of first response of CR or PR, if CR not achieved during follow-up. CR: disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures <10 mm; PR: >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions. Alive participants with no events were censored at date of last response assessment. Data is also presented by de novo status and relapse status.
Time Frame: From index date till first documented CR or PR or date of censoring (for a maximum period of 3 years)
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Palbociclib
Number analyzed (Participants) | 80
Days
  Overall | 115.5 [4.0 to 724.0]
  De novo status: Metastatic disease: number analyzed (Participants) | 28
  De novo status: Metastatic disease | 93.0 [4.0 to 599.0]
  De novo status: Recurrent disease: number analyzed (Participants) | 52
  De novo status: Recurrent disease | 127.5 [53.0 to 724.0]
  Relapse status: More than 12 months: number analyzed (Participants) | 23
  Relapse status: More than 12 months | 105.0 [63.0 to 706.0]
  Relapse status: De novo metastatic disease: number analyzed (Participants) | 28
  Relapse status: De novo metastatic disease | 93.0 [4.0 to 599.0]
  Relapse status: <=12 months: number analyzed (Participants) | 21
  Relapse status: <=12 months | 166.0 [76.0 to 724.0]
  Relapse status: Missing: number analyzed (Participants) | 8
  Relapse status: Missing | 116.0 [53.0 to 258.0]

63. Secondary Outcome: Percentage of Participants With Neutropenia Post-Palbociclib Initiation
Description: Neutropenia is an abnormally low level of neutrophils with count <1500 neutrophils per microliter (mcL) in blood and was classified as per Common Toxicity Criteria (CTC) version 2.0 criteria: grade 1 (mild) with an absolute neutrophil count (ANC) of >=1500 to <2000 cells per mcL, grade 2 (moderate) with an ANC of >=1000 to <1500 cells per mcL, grade 3 (severe) with an ANC of >=500 to <1000 cells per mcL or grade 4 (severe) with an ANC lower than 500 cells per mcL. Percentage of participants with all grades, grade 3 and grade 4 were reported in this outcome measure. All grades category included grades 1 to grade 4.
Time Frame: Data collected from index date up to 6 months post-palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  All grades | 88
  Grade 3 | 40
  Grade 4 | 7

64. Secondary Outcome: Percentage of Participants With Neutropenia Post-Palbociclib Initiation as Recorded and Inferred From Clinical Notes
Description: Neutropenia is an abnormally low level of neutrophils with count <1500 neutrophils per mcL in blood and was classified as per CTC version 2.0 criteria: grade 1 (mild) with an ANC of >=1500 to <2000 cells per mcL, grade 2 (moderate) with an ANC of >=1000 to <1500 cells per mcL, grade 3 (severe) with an ANC of >=500 to <1000 cells per mcL or grade 4 (severe) with an ANC lower than 500 cells per mcL.
Time Frame: Data collected from index date up to 6 months post-palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 190
Percentage of participants
  Grade 1 | 11
  Grade 2 | 14
  Grade 3 | 25
  Grade 4 | 3

65. Secondary Outcome: Percentage of Participants With Neutropenia Post-Palbociclib Initiation as Recorded and Inferred From ANC Measurements
Description: as for outcome 64
Time Frame: Data collected from index date up to 6 months post-palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Grade 1 | 10
  Grade 2 | 31
  Grade 3 | 40
  Grade 4 | 7

66. Secondary Outcome: Percentage of Participants According to the Severe Grade of Neutropenia
Description: Neutropenia is an abnormally low level of neutrophils with count <1500 neutrophils per mcL in blood and was classified as per CTC version 2.0 criteria: grade 1 (mild) with an ANC of >=1500 to <2000 cells per mcL, grade 2 (moderate) with an ANC of >=1000 to <1500 cells per mcL, grade 3 (severe) with an ANC of >=500 to <1000 cells per mcL or grade 4 (severe) with an ANC lower than 500 cells per mcL. Percentage of participants with grade 3 and 4 were reported in this outcome measure.
Time Frame: Data collected from index date up to 3 months post-palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Grade 3 | 37
  Grade 4 | 6

67. Secondary Outcome: Percentage of Participants With Febrile Neutropenia Post-Palbociclib Initiation
Description: Febrile neutropenia (FN) was defined as an ANC of < 1.0 x 10^9 cells/L predicted to fall below 0.5 x 10^9 cells/L within 48 hours with fever or clinical signs of sepsis; fever and ANC were measured the same day or within ± 1 calendar day.
Time Frame: Data collected from index date up to 3 months post-palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 3

68. Secondary Outcome: Percentage of Participants With Gastro-Intestinal Toxicities Post-Palbociclib Initiation
Description: Percentage of participants with gastro-intestinal toxicities as diarrhea, nausea and vomiting after index date were reported in this outcome measure. As per CTC version 2.0 criteria, for diarrhea: grade 1 (mild)- less than 4 stools per day, grade 2 (moderate)- 4 to 6 stools per day, grade 3 (severe)- >=7 stools per day and grade 4 (life-threatening)- physiologic consequences requiring intensive care; Vomiting: grade 1 (mild)- 1 episode per day , grade 2 (moderate)- 2 to 5 episodes per day, grade 3 (severe)- >=6 episodes per day and grade 4 (life-threatening)- physiologic consequences requiring intensive care; Nausea: grade 1 (mild)- able to eat, grade 2 (moderate)- oral intake significantly reduced, grade 3 (severe)- no significant intake and requiring intravenous fluids.
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Diarrhea: All grades | 16
  Diarrhea: Grade 3 | 1
  Diarrhea: Grade not available | 5
  Nausea: All grades | 18
  Nausea: Grade 1 | 12
  Nausea: Grade 2 | 1
  Nausea: Grade not available | 5
  Vomiting: All grades | 11
  Vomiting: Grade 1 | 6
  Vomiting: Grade 2 | 1
  Vomiting: Grade not available | 4

69. Secondary Outcome: Percentage of Participants With Adverse Events During Follow-up
Description: Percentage of participants with at least one of the adverse events (neutropenia, diarrhea, nausea, and vomiting) after index date were reported in this outcome measure.
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants | 72

70. Secondary Outcome: Absolute Values for Hematology Parameter in First 6 Months Following Palbociclib Initiation: Hemoglobin
Description: Absolute values for hematology parameter- hemoglobin, were reported in this outcome measure.
Time Frame: From index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Palbociclib
Number analyzed (Participants) | 183
Grams per liter | 120.5 (10)

71. Secondary Outcome: Absolute Values for Hematology Parameters in First 6 Months Following Palbociclib Initiation: White Blood Cell, Absolute Neutrophil Counts and Platelet Counts
Description: Absolute values for hematology parameters- white blood cell (WBC) counts, absolute neutrophil counts (ANC) and platelet counts (PLT), were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Palbociclib
Number analyzed (Participants) | 183
10^9 cells per liter
  WBC | 4 (1.5)
  ANC: number analyzed (Participants) | 176
  ANC | 2 (1.2)
  PLT | 233.6 (63.8)

72. Secondary Outcome: Absolute Values for Liver Function Parameters in First 6 Months Following Palbociclib Initiation: Aspartate Aminotransferase, Alanine Aminotransferase and Alkaline Phosphatase
Description: Absolute values for liver function parameters- Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase (ALP), were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Palbociclib
Number analyzed (Participants) | 174
International units per liter
  AST: number analyzed (Participants) | 112
  AST | 26.9 (17.9)
  ALT: number analyzed (Participants) | 138
  ALT | 24.5 (19.4)
  ALP | 100.8 (69.3)

73. Secondary Outcome: Absolute Values for Liver Function Parameter in First 6 Months Following Palbociclib Initiation: Albumin
Description: Absolute values for liver function parameter- albumin, were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Palbociclib
Number analyzed (Participants) | 178
Grams per deciliter | 42.8 (4.7)

74. Secondary Outcome: Absolute Values for Liver Function Parameter in First 6 Months Following Palbociclib Initiation: Bilirubin
Description: Absolute values for liver function parameter- bilirubin, were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | Palbociclib
Number analyzed (Participants) | 175
Milligrams per deciliter | 6.9 (3.6)

75. Secondary Outcome: Absolute Values for Bone Profile Parameters in First 6 Months Following Palbociclib Initiation: Calcium and Phosphate
Description: Absolute values for bone profile parameters- calcium and phosphate were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Palbociclib
Number analyzed (Participants) | 167
Millimoles per liter
  Calcium | 2.3 (0.1)
  Phosphate: number analyzed (Participants) | 156
  Phosphate | 1.1 (0.2)

76. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters in First 6 Months Following Palbociclib Initiation: Potassium, Sodium and Urea
Description: Absolute values for clinical chemistry parameters- potassium, sodium and urea were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Palbociclib
Number analyzed (Participants) | 168
Millimoles per liter
  Potassium | 4.3 (0.4)
  Sodium | 139.4 (10.6)
  Urea: number analyzed (Participants) | 152
  Urea | 5.8 (11.2)

77. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter in First 6 Months Following Palbociclib Initiation: Creatinine
Description: Absolute values for clinical chemistry parameter- creatinine, were reported in this outcome measure.
Time Frame: Data collected from index date up to 6 months after palbociclib initiation (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Palbociclib
Number analyzed (Participants) | 168
Micromoles per liter | 70.6 (16.1)

78. Secondary Outcome: Percentage of Participants With Inpatient Admissions and Outpatient Visits
Description: Percentage of participants with inpatient admissions and outpatient visits were reported in this outcome measure.
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  Inpatient Admissions | 28
  Outpatient Visits | 77

79. Secondary Outcome: Number of Inpatient Admissions Per Participant
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Admissions per participant
Arm/Group | Palbociclib
Number analyzed (Participants) | 53
Admissions per participant | 1.4 (0.7)

80. Secondary Outcome: Number of Outpatient Visits Per Participant
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Visits per participant
Arm/Group | Palbociclib
Number analyzed (Participants) | 147
Visits per participant | 9.5 (7.5)

81. Secondary Outcome: Percentage of Participants With Type of Hospital Admission
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 73
Percentage of participants
  Accident and emergency | 86
  Planned | 14

82. Secondary Outcome: Percentage of Participants With Reasons for Hospital Admission
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure. One participant could have more than 1 reason for hospital admission.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 73
Percentage of participants
  Blood tests | 5
  Breathlessness | 8
  Collapse and transfer to the ward | 1
  Hypocalcemia | 1
  Hypoxia | 1
  Incidental deep vein thrombosis (DVT) | 1
  Palliative Mastectomy | 1
  Pleural Effusion | 1
  Pyrexia | 1
  Sepsis | 1
  Shortness of breath and clinically progressive disease | 1
  Small bowel obstruction: no clear cause | 1
  Surgery: appendicectomy | 1
  Swollen/Painful left arm seen by general practitioner (GP)/DVT/cellulitis | 1
  Temperature | 1
  Transfusion | 1
  Unwell | 1
  Urgent review | 66

83. Secondary Outcome: Duration of Inpatient Hospital Stay
Description: Duration of hospital stay was the time from the date of hospital entry to date of hospital discharge.
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Palbociclib
Number analyzed (Participants) | 67
Days | 3 [1.0 to 54.0]

84. Secondary Outcome: Reasons of Outpatient Visit
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, one participant could have more than one event.
Measure: Number; unit: Events
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Events
  Bloods | 40
  Bloods, Zoladex and Denosumab | 3
  Capecitabine pick up | 1
  Chemotherapy | 44
  Dalteparin administration | 1
  Denosumab | 27
  Denosumab + bloods | 2
  Denosumab + Palbociclib handout | 1
  Discontinuation of palbociclib discussed | 1
  Follow-up | 1041
  Genetics testing | 2
  Given treatment | 5
  Goserelin + Denosumab | 1
  Goserelin treatment | 21
  Home visit from palliative care | 3
  Information about disease/treatment | 123
  Insertion of central venous access device | 1
  Lymphoedema review | 2
  Medical concerns | 12
  Oral chemotherapy clinic | 22
  Palbociclib pick up, Zoladex and Denosumab | 9
  Palbociclib Initiation | 2
  Palliative care appointment | 6
  Peripherally inserted central catheter (PICC) line insertion | 2
  Pick up Cyclophosphamide /Methotrexate | 2
  Pick up palbociclib | 3
  Radiotherapy appointment | 1
  Review before discharge | 1
  Treatment initiation | 1
  Trial initiation (1st dose & consent) | 1
  Zoledronic acid | 13

85. Secondary Outcome: Type of Health Care Professional Consultations During Outpatient Visit
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, one participant could consult more than one health care professional.
Measure: Number; unit: Consultations
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Consultations
  Advanced nurse practitioner (ANP) | 47
  Consultant | 772
  Nurse | 284
  Pharmacist | 7
  Specialist registrar (SpR) | 209
  Other | 45
  Not known | 30

86. Secondary Outcome: Percentage of Participants Contacted Cancer National Service (CNS) and Acute Oncology Service (AOS) During First Year After Palbociclib Initiation
Description: Percentage of participants who contacted CNS by phone calls and AOS either by phone calls or visits were reported in this outcome measure.
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Percentage of participants
  CNS | 36
  AOS | 19

87. Secondary Outcome: Percentage of Participants According to Number of CNS Interactions
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 69
Percentage of participants
  1 | 17
  2 | 26
  3 | 19
  4 | 13
  5 | 1
  6 | 4
  7 | 1
  8 | 7
  9 | 4
  10 | 3
  11 | 1
  14 | 1

88. Secondary Outcome: Number of AOS Interactions Per Participant
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Interactions per participant
Arm/Group | Palbociclib
Number analyzed (Participants) | 36
Interactions per participant | 2.1 (1.2)

89. Secondary Outcome: Type of CNS and AOS Interactions
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: FAS comprised of medical records extracted for the purpose of the study from all eligible participants who were enrolled into the study. Here, one participant could have more than one interaction.
Measure: Number; unit: Interactions
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Interactions
  CNS interactions: Phone call | 124
  CNS interactions: Visit | 133
  CNS interactions: Other | 8
  AOS interactions: Phone call | 49
  AOS interactions: Visit | 25

90. Secondary Outcome: Reasons for CNS and AOS Interaction
Time Frame: Data collected from index date up to 1-year of follow up period (for a maximum period of 3 years)
Population: as for outcome 84
Measure: Number; unit: Events
Arm/Group | Palbociclib
Number analyzed (Participants) | 191
Events
  CNS interactions: Follow-up | 157
  CNS interactions: General health and wellbeing check | 2
  CNS interactions: Information about scans/appointments | 2
  CNS interactions: Information about disease/treatment | 44
  CNS interactions: Medical concerns | 44
  CNS interactions: Psychological support | 8
  CNS interactions: Admin issue | 1
  CNS interactions: Clinical letter query | 1
  CNS interactions: Computed tomographic of chest, abdomen and pelvis (CT CAP) query | 1
  CNS interactions: Discussion about further dental work and denosumab injection | 1
  CNS interactions: Not known | 1
  CNS interactions: Pain issues | 1
  CNS interactions: Scan/blood test | 1
  CNS interactions: Treatment schedule | 1
  AOS interactions: Follow-up | 9
  AOS interactions: Information about disease/treatment | 4
  AOS interactions: Inpatient admission | 1
  AOS interactions: Medical concerns | 60

ADVERSE EVENTS:
Time Frame: From baseline up to maximum period of 3 years
Description: Same event may appear as both AE and SAE. But what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or participant may have both serious and non-serious event. AEs were reported as per participants' medical records. There was no specific medical dictionary. 6 participants had febrile neutropenia which was not recorded as SAE or non-SAE as associated grades were not collected as part of electronic case report form (eCRF).
Arm/Group | Palbociclib
All-Cause Mortality (participants affected / at risk) | 3/191
Serious Adverse Events (participants affected / at risk) | 54/191
Other Adverse Events (participants affected / at risk) | 116/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib (N=191)
Neutropenia (Blood and lymphatic system disorders) | 53
Diarrhoea (Gastrointestinal disorders) | 1
Other (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib (N=191)
Neutropenia (Blood and lymphatic system disorders) | 90
Diarrhoea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 24
Other (Gastrointestinal disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03921866/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT03921866/SAP_001.pdf